CLINICAL TRIAL: NCT04608487
Title: A Phase I Study of Anti-CD19 CAR T-cell Therapy With Axicabtagene Ciloleucel (Axi-cel) in Patients With Relapsed/Refractory Primary and Secondary Central Nervous System (CNS) Lymphoma
Brief Title: Axi-cel in CNS Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Kite, A Gilead Company (Industry)
Responsible Party: Principal Investigator, Caron A. Jacobson, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-274
Record Dates: First submitted 2020-10-19; First posted 2020-10-29 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Lymphoma; Lymphoma Cns
Keywords: relapsed/refractory central nervous system (CNS) lymphoma; systemic lymphoma with concurrent CNS lymphoma; systemic lymphoma with a history of treated CNS lymphoma
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; axicabtagene ciloleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fludarabine + Cyclophosphamide + Axicabtagene Ciloleucel (Experimental): Prior to receiving axi-cel, participants will undergo leukapheresis and the need for a Ommaya reservoir placement will be assessed and administered.
  Day -5 to Day -3 of 28 day study cycle Fludarabine and cyclophosphamide; Day -1 admitted to hospital, receive axi-cel on day 0; Till at least cycle day 7 hospital monitoring; post treatment follow up will occur on day 14 and day 28 of cycle 1, monthly in cycles 2, 3, 6, 9,12,15,18,21,24, then yearly after cycle 24.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Axicabtagene Ciloleucel

INTERVENTIONS:
Drug: Fludarabine — Intravenous infusion
  Other Names: Fludara
Drug: Cyclophosphamide — Intravenous infusion
  Other Names: Cytoxan; Neosar
Biological: Axicabtagene Ciloleucel — Intravenous infusion
  Other Names: Yescarta

SUMMARY:
This research is being done to test the safety and effectiveness of axicabtagene ciloleucel (axi-cel), an anti-CD19 directed chimeric antigen receptor (CAR) T-cell therapy in treating relapsed/refractory central nervous system (CNS) lymphoma, systemic lymphoma with concurrent CNS lymphoma, or systemic lymphoma with a history of treated CNS lymphoma, and to better understand what causes neurological toxicity following treatment with axi-cel.

The names of the study drug(s) involved in this study are:

* axicabtagene ciloleucel (axi-cel)
* ludarabine will be given with axicel to help axicel work more effectively
* cyclophosphamide will be given with axicel to help axicel work more effectively

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied. This study will examine the safety and efficacy of axi-cel in participants who either currently or previously had had central nervous system involvement of their lymphoma.

The name of the study drug involved in this study is axi-cel. Axi-cel is a chimeric antigen receptor (CAR) T-cell therapy that is manufactured using a person's own white blood cells. A virus is used to introduce a gene that creates a protein (called a CAR) on the surface of T cells, a type of blood cell that fights infection and can eliminate cancer cells. The CAR on the T cells may bind to and kill cells that express CD19, a molecule that is found on B-cell lymphomas. CAR-T cells (including axi-cel) designed to target CD19, a protein present on B lymphocytes have been used to treat patients with CD19+ tumors. This adoptive cell therapy (ACT) approach has shown significant and durable clinical benefits in the treatment of CD19+ tumors. Axi-cel has been FDA approved for the treatment of relapsed and refractory aggressive B cell lymphomas that occur outside the central nervous system and have recurred after two or more prior therapies.

Participants will receive two chemotherapy medicines, fludarabine and cyclophosphamide. These drugs are not intended as direct cancer treatment but instead to help axi-cel work with less interference from immune system cells.

The research study procedures include screening for eligibility and study treatment including leukapheresis, evaluations and follow up visits.

Participants will receive study treatment once and will be followed for up to 15 years.

It is expected that about 18 people will take part in this research study.

Kite Pharma, a pharmaceutical company, is supporting this research study by providing axi-cel.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed/refractory active primary or secondary CNS lymphoma, histologically proven aggressive B cell lymphoma, including DLBCL, HGBL, PMBL, or tFL, and defined by the following categories:

  * Primary CNS lymphoma, relapsed or refractory following at least one line of CNS-directed therapy. There is no restriction on the number of recurrences.
  * Secondary CNS lymphoma, relapsed or refractory following at least one line of CNS-directed therapy for prophylaxis or treatment of CNS lymphoma.
  * Radiographically event CNS disease by MRI of the brain (ie enhancing lesion on gadolinium enhanced MRI)
  * For patients with secondary CNSL with concurrent systemic lymphoma, the concurrent systemic lymphoma must be either DLBCL, PMBL, high grade B cell lymphoma, or transformed lymphoma and must have relapsed following at least 1 prior lines of therapy (which must have included an anti-CD20 monoclonal antibody (unless the tumor is CD20 negative) and an anthracycline
* At least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic cancer therapy at the time the subject provides consent
* Age 18 years or older at the time of informed consent
* ECOG performance status of 0 or 1
* Adequate bone marrow, renal, hepatic, pulmonary and cardiac function defined as:

  * Absolute neutrophil count (ANC) ≥1000/μL
  * Platelet count ≥ 75,000/μL
  * Absolute lymphocyte count ≥ 100/μL
  * Creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 mL/min
  * Serum alanine aminotransferase/aspartate aminotransferase (ALT/AST) ≤ 2.5 upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5 mg/dl, except in subjects with Gilbert's syndrome
  * Cardiac ejection fraction ≥ 50%, no clinically significant pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings
  * No clinically significant pleural effusion
  * Baseline oxygen saturation > 92% on room air GCSF and transfusions are not allowed for eligibility determination.+++
* Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential)

Exclusion Criteria:

* Primary vitreoretinal lymphoma and intraocular PCNSL without evidence of brain disease. Patients with prior history of intraocular involvement treated only with intraocular methotrexate and no prior systemic therapy are excluded
* PCNSL patients who cannot undergo magnetic resonance imaging assessments
* Patients with brain stem lesions
* Patients with leptomeningeal disease only without brain parenchymal involvement
* Bulky leptomeningeal disease and or CSF protein ≥100 mg/dL
* History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (eg cervix, bladder, breast) unless disease free for at least 3 years
* History of Richter's transformation of CLL
* History of allogeneic stem cell transplant
* Prior CD19 targeted therapy
* Treatment with systemic immunostimulatory agents (including but not limited to interferon and IL-2) within 6 weeks or 5 half-lives of the drug, whichever is shorter, prior to the first dose of axicabtagene ciloleucel or SOC
* Prior chimeric antigen receptor therapy or other genetically modified T-cell therapy
* History of severe, immediate hypersensitivity reaction attributed to aminoglycosides
* Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management. Simple urinary tract infection (UTI) and uncomplicated bacterial pharyngitis are permitted if responding to active treatment.
* Known history of infection with human immunodeficiency virus (HIV) or hepatitis B (HBsAg positive) or hepatitis C virus (anti-HCV positive). If there is a positive history of treated hepatitis B or hepatitis C, the viral load must be undetectable per quantitative polymerase chain reaction (PCR) and/or nucleic acid testing.
* Active tuberculosis
* History or presence of non-malignant CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
* Subjects with cardiac atrial or cardiac ventricular lymphoma involvement
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, New York Heart Association Class II or greater congestive heart failure, or other clinically significant cardiac disease within 12 months of enrollment
* Requirement for urgent therapy due to tumor mass effects
* History of autoimmune disease, requiring systemic immunosuppression and/or systemic disease modifying agents within the last 12 months.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (eg, bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis per chest computed tomography (CT) scan at screening. History of radiation pneumonitis in the radiation field (fibrosis) is allowed.
* History of symptomatic deep vein thrombosis or pulmonary embolism requiring ongoing systemic anticoagulation
* Any medical condition likely to interfere with assessment of safety or efficacy of study treatment
* History of severe immediate hypersensitivity reaction to tocilizumab or any of the agents used in this study
* Treatment with a live, attenuated vaccine within 6 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during the course of the study
* Women of childbearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of chemotherapy on the fetus or infant. Subjects of either sex who are not willing to practice birth control from the time of consent and at least 6 months after the last dose of axicabtagene ciloleucel or SOC chemotherapy
* In the investigators judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2025-06-14 (Actual); Study Completion 2038-06-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE Version 5.0 | Enrollment until 30 days after last dose of study treatment up to 24 Months
  Measured by the rate of TLTs and the rate of grade 3+ adverse events (AEs) regardless of attribution

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  CNS lymphoma response assessment will be evaluated by International Primary CNS Lymphoma Collaborative Group (IPCG) criteria Systemic lymphoma response assessment will be evaluated by the Lugano 2014 criteria
Complete response (CR) rate | 2 years
  CNS lymphoma response assessment will be evaluated by International Primary CNS Lymphoma Collaborative Group (IPCG) criteria Systemic lymphoma response assessment will be evaluated by the Lugano 2014 criteria
Duration of response (DOR) | 2 years
  CNS lymphoma response assessment will be evaluated by International Primary CNS Lymphoma Collaborative Group (IPCG) criteria Systemic lymphoma response assessment will be evaluated by the Lugano 2014 criteria
Progression-free survival (PFS) | 2 years
  CNS lymphoma response assessment will be evaluated by International Primary CNS Lymphoma Collaborative Group (IPCG) criteria Systemic lymphoma response assessment will be evaluated by the Lugano 2014 criteria
Overall survival (OS) | 2 years
  CNS lymphoma response assessment will be evaluated by International Primary CNS Lymphoma Collaborative Group (IPCG) criteria Systemic lymphoma response assessment will be evaluated by the Lugano 2014 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Caron Jacobson, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: the Sponsor Investigator, Dr. Caron Jacobson. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu